CLINICAL TRIAL: NCT06582017
Title: A First-in-human Phase 1a/1b Study to Evaluate Safety and Tolerability of QXL138AM in Patients With Locally Advanced Un-resectable and/or Metastatic Solid Tumors and Multiple Myeloma
Brief Title: Safety, PK and Efficacy of QXL138AM in Patients With Solid Tumors and Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nammi Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QXL138AM-001
Record Dates: First submitted 2024-08-23; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Pancreas Cancer; Urothelial Carcinoma; Renal Cell Carcinoma; Hepatocellular Carcinoma; Gastrointestinal Cancer; Lung Cancer; Prostate Cancer; Breast Cancer
Keywords: QXL138AM-001; CD138; Interferon A; Nammi Therapeutics Inc.
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Gastrointestinal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Modified 3+3 design
Masking Description: Open-label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a Dose Escalation in Solid Tumors - Part A1 (Experimental): Dose escalation of QXL138AM in participants with locally advanced un-resectable and/or metastatic solid tumors.
  Interventions: Biological: QXL138AM Injection every 2 weeks by IV Infusion
- Phase 1a Dose Escalation in Multiple Myeloma - Part A2 (Experimental): Dose escalation of QXL138AM in participants with multiple myeloma.
  Interventions: Biological: QXL138AM Injection every 2 weeks by IV Infusion
- Phase 1b Dose Expansion in Solid Tumors - Part B1 (Experimental): Dose expansion in solid tumors using the recommended dose for expansion from Part A1
  Interventions: Biological: QXL138AM Injection every 2 weeks by IV Infusion
- Phase 1b Dose Expansion in Multiple Myeloma - Part B2 (Experimental): Dose expansion in Multiple Myeloma using the recommended dose for expansion from Part A2
  Interventions: Biological: QXL138AM Injection every 2 weeks by IV Infusion

INTERVENTIONS:
Biological: QXL138AM Injection every 2 weeks by IV Infusion — masked immuno-cytokine comprised of an anti-CD138 IgG1 antibody fused to human interferon alpha 2a

SUMMARY:
Study QXL138AM-001 is a Phase 1a/1b study to investigate the safety, pharmacokinetics, and preliminary activity of QXL138AM in subjects with locally advanced un-resectable and/or metastatic solid tumors and multiple myeloma. The study is an open-label, multicenter, first in human study to be conducted in two major parts which are further organized into two sub-parts. Part A Dose Escalation is a modified 3+3 with the first two cohorts consisting of one subject each based on the low clinical starting dose. Dose escalation in solid tumors (Part A1) will be followed by dose finding in multiple myeloma (Part A2). Part B consists of dose expansion in solid tumors (Part B1) and multiple myeloma (Part B2) using the recommended dose for expansion from Part A

DETAILED DESCRIPTION:
This is an open-label, multicenter, first in human (FIH) Phase 1a/1b study of QXL138AM in participants with locally advanced unresectable and/or metastatic solid tumors and multiple myeloma. This study will be conducted in two parts (A and B) and each part has two sub-parts for tumor type (1 and 2).

Part A1 - Dose Escalation in Solid Tumors The following solid tumor types will initially be enrolled in this part: ovarian, pancreatic, urothelial, renal, hepatocellular, gastrointestinal, lung, prostate, and breast cancer.

Dose escalation will use a standard 3+3 design, where 3 to 6 participants with advanced solid tumors will be enrolled sequentially into each cohort/dose level with the exception of Cohort 1 and 2. For Cohorts 1 and 2, given the very low starting dose, only one participant is planned for each level unless a participant experiences a Grade 2 or higher adverse event not clearly and incontrovertibly related to disease progression or an extraneous factor. If such a Grade 2 or higher event occurs in Cohort 1 or 2, dose escalation will switch to a standard 3+3 design. Dose escalation will continue until the MTD or RDE is determined in participants with solid tumors, referred to as the RDE-ST. At this point, the two solid tumor types for dose expansion will be selected for Part B1 and may begin at the RDE-ST.

The proposed dose levels are defined in the table below. Cohort No. of Participants Dose Level (Q2W) (mg/kg)

1. 1-6 0.001
2. 1-6 0.003
3. 3-6 0.01
4. 3-6 0.03
5. 3-6 0.1
6. 3-6 0.3
7. 3-6 1
8. 3-6 2
9. 3-6 4 Infusions will be administered via syringe pump or IV bag (depending on the dose) and administered over a 30-60-minute (± 10 minutes) duration.

Part A2 - Dose Escalation in Multiple Myeloma Dose escalation in multiple myeloma will commence when the RDE-ST for solid tumors has been identified, or if there are signs of anti-tumor activity in Part A1 as determined by the Sponsor.

Dose escalation will use a standard 3+3 design, where 3 to 6 participants with multiple myeloma will be enrolled sequentially into dose escalation cohorts starting at one dose level below the RDE-ST determined from solid tumor dose escalation (RDE-ST-1). Alternatively, if signs of anti-tumor activity in Part A1 are observed, the Sponsor may elect to initiate dose escalation in multiple myeloma at one dose level below the highest dose already deemed safe in Part A1. If two of the first six participants in the first multiple myeloma cohort experience a DLT, then the dose will be further reduced by one level (RDE-ST-2). Once the RDE for multiple myeloma patients is determined, it will be referred to as the RDE-MM and dose expansion may begin in patients with multiple myeloma at this dose.

Part B1: Dose Expansion in Solid Tumors When the RDE-ST has been identified by the SRC from Part A1, the study may continue to Part B1 dose expansion to further explore the safety and anti-tumor activity of QXL138AM in solid tumors. Dose expansion will enroll two cohorts of 20 participants each in two solid tumor indications identified from Part A1. In each cohort, patients will be randomized 1:1 to receive the RDE-ST dose or 1 dose lower. The Sponsor may opt to enroll additional participants up to a maximum of 40 in each cohort if signs of anti-tumor activity are observed.

Part B2: Dose Expansion in Multiple Myeloma When the RDE-MM in multiple myeloma has been identified by the SRC from Part A2, the study may continue to Part B2 dose expansion to further explore the safety and anti-tumor activity of QXL138AM in patients with multiple myeloma. Up to 20 participants will be treated at the RDE-MM identified in Part A2. Patients will be randomized 1:1 to receive the RDE-MM dose or 1 dose lower.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Solid Tumors

   * Histopathologically confirmed diagnosis of an advanced, unresectable, or metastatic solid tumor (ovarian, pancreatic, urothelial, renal, hepatocellular, gastrointestinal (GI), lung, prostate, and breast cancer).
   * Have progressed despite standard therapies, or for whom conventional therapy is not effective or tolerable, as judged by the Investigator. Patients must have no available therapeutic options known to confer clinical benefit for their tumor type.
2. Participants with Multiple Myeloma

   * Have progressed despite standard therapies, or for whom conventional therapy is not effective or tolerable, as judged by the Investigator.
   * Patients must have failed at least 3 prior therapies for myeloma and should have had prior exposure to a proteosome inhibitor, an IMiD, and an anti-CD38-directed therapy.

2. Male or female participants ≥18 years of age at the time of informed consent 3. An Eastern Cooperative Oncology Group (ECOG) performance status scale of 0, 1, or 2 at Screening 4. Must have at least 1 measurable lesion by RECIST version 1.1 (solid tumors only), or evaluable disease by IMWG Uniform Response Criteria (multiple myeloma only) 5. Adequate organ function and bone marrow reserve 6. Adequate cardiac function as estimated by left ventricular ejection fraction 7. Female participants of child-bearing potential must:

* Have a negative serum pregnancy test at screening and a negative pregnancy test at Week 1 Day 1 prior to first dose of QXL138AM, AND
* Agree to use at least 1 highly effective method of contraception for the duration of study participation, and for 120 days after last dose of QXL138AM.

  8. Male participants of child-bearing potential must:
* Agree to use at least 1 highly effective method of contraception for the duration of study participation, and for 120 days after last dose of QXL138AM, AND
* Refrain from sperm donation prior to the first dose of investigational product through 120 days following the last dose of QXL138AM.

Exclusion Criteria:

1. New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, a history of risk factors for Torsades de Pointes (TdP), including heart failure, hypokalemia, and family history of long QTc syndrome, or evidence of ischemia on ECG.

   Symptomatic ischemic heart disease or unstable angina pectoris; or history of cardiac angioplasty, cardiac stenting, or coronary artery bypass graft. A clinically significant baseline prolongation of QT/QTcF interval at screening.
2. The use of concomitant medications that may significantly prolong the QT/QTc interval.
3. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
4. Known hypersensitivity to the investigational product or components (anti-CD138 IgG1 antibody, Interferon A2a and/or the formulation excipients: histidine, sucrose, arginine, polysorbate 80).
5. Female participant is lactating.
6. Any other clinically significant comorbidities.
7. Received prior anticancer therapy within 28 days or 5x the half-life (whichever is shorter) prior to the first dose of investigational product.
8. Participants who received wide-field radiation therapy within 4 weeks prior to first dose of investigational product, (2 weeks for limited field radiation therapy)
9. Major surgery within 30 days before first dose of investigational product
10. Chronic use of systemic corticosteroids of more than 20 mg/day of prednisone or equivalent.
11. Active, clinically significant liver disease such as Hepatitis B or C, autoimmune hepatitis, or cirrhosis (Child Hugh Stage B or C).
12. Current or history of mood disorder such as major depression per DSM-5 within past two years not controlled with current therapy.
13. Active autoimmune disorders not controlled with current therapy.
14. Active endocrine disorders including hypothyroidism, hyperthyroidism, hypoglycemia, hyperglycemia, and diabetes mellitus not controlled with current therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Throughout study - anticipated 3.5 years
  Record all safety events during study including AEs, SAEs, DLTs, AESIs.

SECONDARY OUTCOMES:
Measurement of maximum plasma concentration (Cmax) of QXL138AM | Throughout study - anticipated 3.5 years
  Measured from blood samples
Describe Anti-tumor activity | Part B of study - anticipated 1.5 years
  Indices of anti-tumor activity (using RECIST 1.1 for solid tumors) and International Myeloma Working Group [IMWG] Uniform Response Criteria for multiple myeloma) such as overall response rate (ORR), progression-free survival (PFS), time to response (TTR), duration of response (DOR), minimal residual disease (MRD) and overall survival (OS) during treatment (Part B only)
Measurement of trough concentration (Ctrough) of QXL138AM | Throughout study - anticipated 3.5 years
  Measured from blood samples
Measurement of area under the serum concentration-time curve (AUC) of QXL138AM | Throughout study - anticipated 3.5 years
  Measured from blood samples
Incidence of Anti-drug Antibodies | Throughout study - anticipated 3.5 years
  Measured from blood samples

OTHER OUTCOMES:
Measurement of Exploratory Biomarkers | Throughout study - anticipated 3.5 years
  Identify any correlation between CD138 expression in tumors and anti-tumor response and to characterize the changes in serum cytokine levels such as: IFN- , TNF-α, IL-6 and IL-2

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD, Study Director — Nammi Therapeutics Inc
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Cedars-Sanai Medical Center - Samuel Oschin Comprehensive Cancer, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport, California
  - Sarah Cannon Research Institute - Denver DDU, Denver, Colorado
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - New York Cancer & Blood Specialists, New York, New York
  - University of Rochester - Wilmot Cancer Institute, Rochester, New York
  - START San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No